CLINICAL TRIAL: NCT03999216
Title: Creating a Platform for Point-of-Care Pragmatic Clinical Trials: Comparing Diuretic Strategies in Heart Failure
Brief Title: Comparing Diuretic Strategies in Hospitalized Heart Failure
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to administrative and logistical barriers this trial has been withdrawn.
Sponsor: Stanford University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Tara I-Hsin Chang, Associate Professor of Medicine (Nephrology), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51720
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
Keywords: diuretics
MeSH Terms: conditions — Heart Failure | interventions — Sodium Chloride Symporter Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loop only (Active Comparator): Participants will receive a loop diuretic for up to the first 72 hours of hospitalization. The specific drug, dose and route are left to the treating providers.
  Interventions: Drug: Loop Diuretics vs. loop + thiazide diuretics
- Loop + Thiazide (Active Comparator): Participants will receive a loop+thiazide diuretic for up to the first 72 hours of hospitalization. The specific drugs, doses and routes are left to the treating providers.
  Interventions: Drug: Loop Diuretics vs. loop + thiazide diuretics

INTERVENTIONS:
Drug: Loop Diuretics vs. loop + thiazide diuretics — Participants will receive the diuretic type as determined by the randomized group assignment starting within the first 24 hours of hospital admission and continuing for up to 72 hours. All other treatments are left to the discretion of the treatment team, as this is a pragmatic randomized trial.

SUMMARY:
We will conduct a pragmatic randomized trial comparing whether using a combination of two types of diuretics (loop + thiazide) compared with using a single diuretic (loop only) will result in shorter hospital stays for patients hospitalized with heart failure.

ELIGIBILITY:
Inclusion Criteria:

Any adult (age ≥18 years) admitted to the Heart Failure Service at Stanford Health Care with an indication for treatment with a diuretic.

Exclusion Criteria:

1. admission to the intensive care unit or cardiac care units
2. maintenance dialysis on admission
3. any mechanical circulatory support on admission
4. history of heart transplant
5. allergy / intolerance to loop or thiazide diuretics
6. admission serum sodium < 125 meq/L (from EPIC)
7. admission serum potassium < 3.0 meq/L (from EPIC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | During hospitalization up to 90 days

SECONDARY OUTCOMES:
Composite of all-cause rehospitalizations, emergency department visits, or death in the 30 days after hospital discharge. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tara Chang, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No